CLINICAL TRIAL: NCT07255066
Title: Optimizing Patient Treatment With EPA-enriched Nutrition, a Randomised Control Trial
Acronym: OPT-EPA
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Edinburgh (Other)
Collaborators: University of Southampton (Other); Danone Global Research & Innovation Center (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AC25085; 2024-07601 (Other Grant/Funding Number: Danone Global Research and Innovation)
Record Dates: First submitted 2025-11-19; First posted 2025-11-28 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Malnutrition (Calorie); Colorectal Cancer; Lung Cancer
MeSH Terms: conditions — Malnutrition; Colorectal Neoplasms; Lung Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dietary Counselling and EPA-enriched FFS (experimental ONS) and standard care (Experimental)
  Interventions: Dietary Supplement: Fortimel Forticare Sensations
- Dietary Counselling and standard care (No Intervention)

INTERVENTIONS:
Dietary Supplement: Fortimel Forticare Sensations — An EPA-enriched experimental Oral Nutritional Supplement
  Arms: Dietary Counselling and EPA-enriched FFS (experimental ONS) and standard care

SUMMARY:
Malnutrition is a common and serious issue for people living with cancer. Many cancer patients experience weight loss, muscle weakness, and poor quality of life due to malnutrition. This can also reduce the success of cancer treatments, increase hospital visits, and add emotional distress for both patients and their loved ones.

Treating malnutrition through good nutritional care is increasingly recognised as an important part of cancer treatment. Leading experts recommend that all cancer patients be checked for signs of malnutrition and given personalised nutrition plans when necessary. While dietary counselling and oral nutritional supplements (ONS) are often used to help patients, there is still a need for better evidence to show how well these interventions work.

A key factor contributing to malnutrition in cancer patients is inflammation. Omega-3 fatty acids, (like those found in oily fish) are known for their anti-inflammatory properties. Some studies suggest that omega-3s may help cancer patients by reducing inflammation, keeping muscles strong, improving appetite, and enhancing overall well-being.

The OPT-EPA study will investigate whether a nutritional drink, called Fortimel Forticare Sensations (FFS), can improve nutritional status in patients with lung or colorectal cancer who are at risk of malnutrition. This drink is enriched with omega-3 fatty acids (Eicosapentanoic acid (EPA) and Docosahexaenoic acid (DHA)) and provides a high amount of protein and calories in a small volume, making it easier to consume, especially for patients with taste changes.

In this study, participants will be divided into two groups. The experimental group will receive dietary counselling and standard care along with FFS, the omega-3-enriched nutritional drink, while the other (control) group will receive dietary counselling and standard care, with supplements provided only if clinically necessary. Researchers will evaluate the impact on patients' nutritional status, body weight, muscle, inflammation levels, and quality of life.

Through the OPT-EPA study, researchers hope to gain clearer insights into whether omega-3-containing supplements can provide meaningful benefits for cancer patients. Ultimately, this could help improve the quality of care and outcomes for people facing cancer-related malnutrition.

ELIGIBILITY:
Inclusion Criteria:

* Participants with stage III-IV lung and/or colorectal cancer undergoing systemic anti-cancer treatment (SACT) or starting SACT within the next 4 weeks *with non-curative intent
* Participants aged 18 or older
* Participants at nutritional risk defined as a BMI <20 kg/m2 and/or weight loss between 5-10% in the previous 6 months**
* Participants with systemic inflammation within 28 days of screening (e.g. CRP >10 mg/dL)
* Participants with an ECOG-PS*** score of 0, 1 or 2
* Participants willing and able to give written informed consent

Exclusion Criteria:

* Participants with a recent history of tumour resection (within 12 months)
* Participants who have lost >10% body weight in the previous 6 months before baseline - observed or participant reported.
* Participants with severe renal or hepatic failure or an intolerance to any of the ingredients of the study product
* Participants who are using dietary counselling, ONS or any form of artificial feeding at the time of recruitment
* Unable to adhere to either arm of the trial and appropriate requirements
* Contraindication to ONS including a lactose intolerance
* Females who are pregnant or of childbearing potential and not using adequate contraception

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 118 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2027-01 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Body Weight - light clothes, no shoes | From baseline to day 56